CLINICAL TRIAL: NCT00376727
Title: A Phase I Study of the Safety and Tolerability of Four Doses of Cetuximab (C225) in Patients With Advanced Solid Tumors
Brief Title: Cetuximab in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Angela Davies, MD, University of California, Davis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000506089; P30CA093373 (NIH); UCDCC-165 (Other: University of California, Davis - Cancer Center); BMS-CA225027 (Other Grant/Funding Number: Bristol-Myers Squibb); 200412499 (Other: University of California, Davis - IRB); IMCL-8420 (Other Grant/Funding Number: Imclone Systems, Inc.)
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Cetuximab; Molecular Diagnostic Techniques; Immunologic Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I dose escalation study (Experimental)
  Interventions: Biological: cetuximab; Genetic: molecular diagnostic method; Other: immunologic technique; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: cetuximab — Dose level 0: cetuximab 400 mg/m2 week 1, 250 mg/m2 weekly; Dose level 1: cetuximab 400 mg/m2 week 1, 300 mg/m2 weekly; Dose level 2: cetuximab 400 mg/m2 week 1, 350 mg/m2 weekly; Dose level 3: cetuximab 400 mg/m2 week 1, 400 mg/m2 weekly
  Other Names: IMC-C225; Erbitux
Genetic: molecular diagnostic method — Tissue and Blood Specimens; IHC Methodology; IHC Scoring; K-RAS Mutation Analysis
Other: immunologic technique — Peripheral Blood Mononuclear Cells (PBMC)
Other: laboratory biomarker analysis — Cetuximab Pharmacodynamics

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This phase I trial is studying the side effects and best dose of cetuximab in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of cetuximab in patients with advanced solid tumors.

Secondary

* Evaluate the safety and tolerability of this drug in these patients.
* Develop a detailed scale for assessment of rash in these patients.
* Investigate potential predictors of response using correlative studies on patient tissue, buccal mucosa, and blood samples.
* Obtain preliminary efficacy data and evaluate the relationship of efficacy to grade of rash.
* Correlate downstream markers (e.g., pMAPK, pAKT, and Ki-67) and the presence of epidermal growth factor receptor (EGFR) polymorphisms with clinical response and/or survival.
* Examine the levels of downstream marker proteins in buccal cells obtained pre- and post-treatment.
* Correlate basal p27 expression levels with response and/or survival.
* Determine if the presence of a K-RAS mutation influences response or survival outcome.
* Correlate the presence or absence of mutant K-RAS tumor DNA shed into patient plasma with response and/or outcome.
* Correlate levels of cytokines and chemokines with rash and clinical response.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive cetuximab IV over 90 minutes once weekly for 4 weeks. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of cetuximab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

Patients undergo blood and buccal mucosa collection at baseline and prior to courses 2 and 3 of treatment for molecular correlative studies. Archival tumor tissue specimens are also used for molecular correlative studies. Immunologic correlative studies are performed using patient blood samples.

After completion of study treatment, patients are followed periodically for survival.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Histologically or cytologically proven advanced solid tumors not curable by surgery, radiation therapy or standard chemo-, immuno-, or hormonal therapy. A specific primary cancer need not have been identified (i.e., unknown primary is eligible).
* Patients must have received at least one prior regimen (chemotherapy and/or radiation) for metastatic disease. There is no limit to the number of prior therapies.
* Any prior chemotherapy must have been completed at least 4 weeks prior to start of study therapy. Previous radiation therapy must have been completed at least 2 weeks prior to start of study therapy. All side effects of prior therapy must be resolved prior to the start of study therapy.
* Patients with ZUBROD performance status 0-2 (see Appendix 1).
* Patients must have measurable disease or evaluable disease.
* Patients must have an estimated survival of at least 3 months.
* Patients with asymptomatic treated brain metastasis (surgical resection or radiotherapy) may be included if they are neurologically stable and have been off steroids for at least 4 weeks.
* Patients >/= 18 years of age.
* Patients of reproductive potential must agree to use an effective contraceptive method while on treatment and for 3 months afterward as the effects of cetuximab on the unborn fetus are unknown.
* Patients must have adequate hematologic function defined as: ANC >/= 1,500/mm3, platelets >/= 100,000/mm3.
* Patients must have adequate hepatic function defined as SGOT </= 3 x institutional UNL and serum bilirubin </= 2.0 mg/dL.
* Patients must have adequate renal function defined as a serum creatinine level </= 1.6 mg/dL or a calculated creatinine clearance of >/= 40 ml/min.

Exclusion Criteria:

* Female patients cannot be pregnant or breastfeeding as the effects of cetuximab on the unborn fetus are unknown. Documentation of a negative pregnancy test prior to treatment is required for all women of reproductive potential.
* Uncontrolled intercurrent illness including but not limited to ongoing infection or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.
* Patients with symptomatic brain metastasis or still requiring steroids.
* Patients who have received prior cetuximab therapy, prior therapy with any other drug that targets the EGF receptor (including, but not limited to, Iressa, Tarceva, Herceptin, CI1033, etc.), or prior therapy with a monoclonal antibody.
* Patients who have received prior chemotherapy within 4 weeks or radiation therapy within 2 weeks prior to the start of study therapy.
* Prior hypersensitivity reaction to chimerized or murine monoclonal antibody therapy.
* Patients may not receive any other chemotherapy, radiation therapy, or biologic therapy while on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2004-12; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of cetuximab | December 2007

SECONDARY OUTCOMES:
Safety and tolerability of cetuximab | December 2007
Potential predictors of response using correlative studies | December 2007
Correlation of efficacy of cetuximab with grade of skin rash | December 2007
Development of a detailed scale for assessing skin rash | December 2007

CONTACTS AND LOCATIONS:
Overall Officials: Angela Davies, MD, Study Chair — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States